CLINICAL TRIAL: NCT02904616
Title: Validation of a Medical Device, a Mobile Spectrofluorimeter, Measuring Skin Autofluorescence in Healthy Volunteers
Acronym: PHOTOFLUO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014-A01220-47
Record Dates: First submitted 2016-09-02; First posted 2016-09-19 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteers (Experimental): Healthy volunteers wash their hands with a traditional soap. Every healthy volunteers pose with palm of hand three times on the device in order to measure basal level of fluorescence of the skin.
  Healthy volunteers repeated three times this procedure in order to assess the reproducibility of the measurement.
  Interventions: Device: mobile spectrofluorimeter

INTERVENTIONS:
Device: mobile spectrofluorimeter

SUMMARY:
The Institut has developed a spectrofluorimeter for the registration and monitoring of skin autofluorescence.

This Spectrofluorometer must be initially validated in healthy volunteers. In the long term, it will be used clinically to measure residual photosensitivity of patients who received a photosensitizer in photodynamic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Man and woman over 18 yers old
* Women of childbearing age under contraceptive
* Healthy volunteers able and willing to follow all procedures of the agreement with the study protocol.
* Healthy volunteers affiliated to the social security
* Ability to provide written informed consent
* Patient's legal capacity to consent to study participation

Exclusion Criteria:

* Healthy volunteers with scars or open wounds on the palms
* Healthy volunteers with warts on their hands
* Healthy volunteers with blister on their hands
* Healthy volunteers involved in another clinical trial
* Pregnant or breastfeeding women
* People in emergencies
* Deprived of liberty or under supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-01-26 (Actual); Primary Completion 2015-02-05 (Actual); Study Completion 2015-02-05 (Actual)

PRIMARY OUTCOMES:
Intraindividual reproducibility of measuring the natural and basal skin fluorescence | 1 day
  The intra-individual reproducibility of measurement of natural and basal skin fluorescence will be evaluated on a healthy volunteers using a mobile spectrofluorimeter. The value of intra-class correlation coefficient will be measured by the method of Fleiss (Fleiss, 1986).

SECONDARY OUTCOMES:
Demographic parameter | 1 day
  gender
Concomitant treatments | 1 day
  Concomitant treatments ( anti-inflammatory antihistaminic, antifungal...) influencing the natural and basal skin fluorescence will be listed.
Dominant hand | 1 day
  left hand / right hand

CONTACTS AND LOCATIONS:
Overall Officials: Guillemin François, MD, PUPH, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No